CLINICAL TRIAL: NCT02380495
Title: Studio NaVA - Studio Nazionale Sulla Qualità Della Vita in Adolescenti Con Rinite Allergica Con e Senza Asma
Brief Title: "Studio NaVA" - National Study on Quality of Life in Adolescents Affected by Allergic Rhinitis With or Without Asthma
Status: Completed | Type: Observational
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Other Study IDs: Verbale n°13/2013
Record Dates: First submitted 2015-02-27; First posted 2015-03-05 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Allergic Rhinitis; Asthma
Keywords: Adolescents; Respiratory Pathology
MeSH Terms: conditions — Rhinitis, Allergic; Asthma | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Allergic rhinitis with/without asthma, from 14 to 17 years age: 600 adolescents with allergic rhinitis with/without asthma, from 14 to 17 years age, recruited from Pediatricians of the Italian territory.
  Interventions: Other: Data Collection
- Without respiratory pathology: 600 subject (5 for each participant Pediatrician) of the same age range, without respiratory pathology (patient family)
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection

SUMMARY:
"Studio Nava" is a National Study aiming to assess allergic rhinitis and asthma outcomes on Quality of Life and Quality of Sleep in adolescent patients by means of Web Survey. "Studio Nava" also proposes the innovative use of a web platform ("http://nava.ibim.cnr.it/") that contains all standardized tools (medical-healthcare web form, ACT, Asthma control test; PSQI, Pittsburgh Sleep Quality Index; T5SS, Total Symptom Score; modified SIDRIA for adolescents; Rhinasthma; VAS scale), that will be available for the doctors after the registration to the web platform. Downloaded questionnaires will be delivered to case-patient, asking him/her to fill them during the waiting time of the visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical cases n°: 600 adolescents affected by allergic rhinitis with/without asthma, from 14 to 17 years age.
* Controls n°: 600 subject (5 for each participant Pediatrician) of the same age range, without respiratory pathology.

Exclusion Criteria:

* Subjects that have not allergic rhinitis with/without asthma diagnosis or are <14 years old or >17 years old

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * 600 adolescents with allergic rhinitis with/without asthma, from 14 to 17 years age, recruited from Pediatricians of the Italian territory
  * 600 subject (5 for each participant Pediatrician) of the same age range, without respiratory pathology (patient family)
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the allergic rhinitis impact on quality of life | 2 weeks

SECONDARY OUTCOMES:
The impact of AR and asthma on quality of sleep | 2 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily
  - Institute of Biomedicine and Molecular Immunology, IBIM, Palermo